CLINICAL TRIAL: NCT07212309
Title: The Effect of a Six-Week Board Game-Based Educational Intervention on Hydration Knowledge, Status, and Practices in Tunisian School Children
Brief Title: Six-Week Board Game Intervention to Improve Hydration in Tunisian School Children
Acronym: HYDRAGAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Higher Institute of Sport and Physical Education of Sfax (Other)
Responsible Party: Principal Investigator, Sana Kacem, Principal Investigator, The Higher Institute of Sport and Physical Education of Sfax
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HydrationBoardGame2021
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Hydration Status; Hydration Behavior; Water Intake
Keywords: hydration; hydration knowledge; water intake; Physical Education; Board Game Intervention

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial with classes assigned as clusters to either the board game educational intervention or the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Board Game-Based Hydration Education (Experimental): Children in this group participate in a six-week educational program using board games designed to improve hydration knowledge, encourage healthy drinking behaviors, and monitor hydration status. Sessions are interactive, engaging, and integrated into school activities
  Interventions: Behavioral: Board Game-Based Hydration Education Program
- Control Group - Usual School Activities (No Intervention): Children in this group continue their usual school routine without any additional educational program on hydration. They serve as a comparison to evaluate the effects of the intervention

INTERVENTIONS:
Behavioral: Board Game-Based Hydration Education Program — A six-week educational program delivered through board games, designed to improve hydration knowledge, practices, and status among school children. The program includes interactive sessions, quizzes, and games that teach the importance of adequate water intake. It is integrated into regular school activities and monitored for engagement and adherence.
  Arms: Intervention Group - Board Game-Based Hydration Education

SUMMARY:
This study evaluated a six-week educational program designed to improve hydration knowledge, hydration status, and drinking practices in young school children in Tunisia. The intervention used an adapted "Snakes and Ladders" board game that delivers fun, age-appropriate messages about healthy fluid intake.

Two hundred forty first-grade students (ages 6-7 years) from two public primary schools were invited to participate during the 2021-2022 academic year. After obtaining parental consent, children were assigned by class to either an intervention group, which played the hydration board game once a week before their physical education (PE) lesson, or a control group, which continued usual activities.

Primary outcomes included hydration knowledge, hydration status (change in body mass before and after PE), perceived thirst, and the volume of water consumed during PE. Outcomes were measured before the program and again after six weeks. This randomized controlled trial sought to determine whether a playful, classroom-based board game can enhance children's understanding and daily practices related to proper hydration.

DETAILED DESCRIPTION:
Adequate hydration is a critical determinant of children's physical health, cognitive functioning, and participation in daily school activities. Despite the well-documented benefits of maintaining optimal hydration, evidence consistently demonstrates that many school-aged children consume insufficient amounts of water during the school day. This inadequacy may compromise physical performance, learning capacity, and general well-being. Consequently, effective and engaging strategies are required to promote hydration-related knowledge and foster sustainable drinking behaviors in school settings.

This study employed a cluster-randomized controlled trial design to evaluate the effectiveness of a six-week board game-based educational intervention in enhancing hydration knowledge, hydration status, and fluid consumption among Tunisian primary school children. The intervention was conceived as an innovative, developmentally appropriate approach that integrates health education within a playful learning format.

Participating schools were randomly allocated at the class level to either the intervention group or the control group. The intervention consisted of weekly sessions in which children played an adapted version of the traditional "Snakes and Ladders" board game. The game was modified to incorporate hydration-related messages: ladders symbolized appropriate hydration practices, while snakes represented missed opportunities to drink water. Each session lasted approximately 30 minutes and was conducted immediately prior to scheduled physical education lessons. Teachers facilitated gameplay, guided discussion, and reinforced key messages. Children assigned to the control group continued their usual educational activities without exposure to the intervention.

Primary outcomes focused on cognitive, behavioral, and physiological aspects of hydration. Specifically, researchers examined changes in children's hydration knowledge, hydration status during physical education, perceived thirst, and water intake across the intervention period. Baseline and post-intervention assessments were conducted to evaluate program impact.

By embedding health-related messages into a culturally adapted, game-based learning tool, this study seeks to assess the feasibility and effectiveness of playful education in fostering positive hydration behaviors. The findings are expected to contribute to the evidence base for innovative school-based health promotion strategies and may provide valuable insights for educators and public health practitioners aiming to enhance children's well-being through accessible, low-cost interventions.

ELIGIBILITY:
Inclusion Criteria:

* First-grade students aged 6-7 years
* Normal BMI according to Cole criteria (2007)
* Parental consent provided

Exclusion Criteria:

* Exempted from PE due to injury, allergy, or medical condition
* Absent during data collection

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in hydration knowledge among school children | From baseline to end of six-week intervention
  Hydration knowledge was assessed using the Hydration Awareness Questionnaire (HAQ), a validated instrument designed to evaluate understanding of hydration concepts, acclimatization, and their importance for safe exercise. The HAQ consists of 15 items, each scored on a 0-10 Likert scale (0 = strongly disagree, 10 = strongly agree), for a total possible score of 0-150, with higher scores indicating greater hydration knowledge. The primary objective is to determine whether the board game-based educational intervention improves children's hydration knowledge relative to the control group.

SECONDARY OUTCOMES:
Change in self-reported hydration habits among school children | Pre- and post-intervention over six weeks
  Self-reported hydration practices were assessed using the Hydration Habits Questionnaire (HHQ), a validated instrument consisting of 7 items. The HHQ evaluates the frequency of fluid intake, type of drinks consumed, source of fluids, and perceived barriers to drinking. Questions are answered using either a 0-10 Likert scale (0 = never, 10 = always) or multiple-choice responses, with some items requiring explanation of the selected response. Higher scores indicate more frequent or better hydration behaviors. This measure evaluates whether children increase water consumption and adopt healthier hydration habits during the intervention.
Hydration status | before and after their PE lesson during six weeks
  determined as the percentage change in body weight before and after their PE lesson.
Change in observed hydration behavior during school physical education sessions | Pre- and post-intervention over six weeks
  Observed hydration behavior was assessed by trained research staff during physical education sessions. The assessment included recording the number of drinking occasions, volume of water consumed (mL), and appropriate use of water breaks. These structured observations were conducted weekly for each child to evaluate whether participation in the board game-based educational program leads to improved hydration practices in the school setting.

CONTACTS AND LOCATIONS:
Locations (1):
- Higher Institute of Sport and Physical Education of Sfax, Tunis, Sfax Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No